CLINICAL TRIAL: NCT01619241
Title: The Role of F-18 FLT PET/CT for Selecting the Patients Who Need Maintenance Treatment After First-line Chemotherapy in Advanced Non-small Cell Lung Cancers
Brief Title: Pilot Study for Evaluating the Role of F-18 FLT PET/CT in Therapeutic Decision Making in Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Ie Ryung Yoo, Chief of Nuclear Medicine department, The Catholic University of Korea
Other Study IDs: KC12EISI0104; KC12EISI0104 (Other: Seoul St.Mary's Hospital Institutional Review Board)
Record Dates: First submitted 2012-05-24; First posted 2012-06-14 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: lung cancer; F-18 FLT PET/CT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- advanced non-small cell lung cancer
  Interventions: Other: PET/CT

INTERVENTIONS:
Other: PET/CT — F-18 FLT PET/CT
  Other Names: F-18 FLT PET/CT

SUMMARY:
The objective of this pilot study is to determine whether 18F-FLT PET/CT can predict which patients will have poorer progression free survival and overall survival in advanced Non-small Cell Lung Cancer (NSCLC) after first-line therapy and, therefore, need more aggressive treatment.

DETAILED DESCRIPTION:
Standard therapy for patients with advanced NSCLC is platinum based doublet chemotherapy. Current first-line chemotherapy is usually limited to 4-6 cycles, as prolonging treatment does not result in additional benefit and may often cause further toxicity. Until recently, treatment guidelines recommended withholding administration of later-line systemic anti-cancer treatment until disease progression.

There are several reports suggesting that maintenance therapy following first-line chemotherapy offers improved survival in advance stage patients. This approach involves the administration of an active treatment immediately after first-line chemotherapy, thus maintaining the clinical benefit initially obtained. However, drug related toxicity and costs are of great concern. There may also be patients with less aggressive disease where an immediate transition to maintenance therapy after first-line results in overtreatment.

Therefore, selecting patients who require more aggressive treatment or earlier intervention is necessary.

If FLT PET/CT can discriminate the patients with shorter progression free survival and overall survival in this pilot study, patients could be selected for more aggressive or earlier treatment such as maintenance therapy, and the investigators could expect to prolong survival while reducing the adverse events and costs that will accompany inconsequential therapy with FLT PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* advanced non-small cell lung cancer (stage IIIB, IV)
* at least one measurable lesion
* performance status (ECOG) 0-2
* 1st-line platinum chemotherapy and no progression

Exclusion Criteria:

* mixed small cell and non-small cell
* uncontrolled brain metastasis
* previous malignancy within 5 years (except basal cell carcinoma of skin, carcinoma in situ of uterine cervix)
* pregnant or breast feeding
* pemetrexed chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advanced non-small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
overall survival | from the date of FLT PET/CT to the date of death or last follow-up, assessed up to 1 year

SECONDARY OUTCOMES:
time to progression | from the date of FLT PET/CT to the date of documented progression or last follow-up, assessed up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ie Ryung Yoo, MD, Principal Investigator — Seoul St. Mary's Hospital; Jin Hyoung Kang, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St.Mary's Hospital, Seoul, South Korea